CLINICAL TRIAL: NCT00521222
Title: Arg/Arg Genotype and Long Acting Beta Agonists in Asthma. Improved Quality of Care for Patients With Asthma.
Brief Title: Evaluating Long Acting Beta Agonists Used to Treat Asthma Among Those With Either Arg/Arg or Gly/Gly Genotypes
Acronym: ARGARG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAC1135
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Asthma
Keywords: asthma; beta agonist; bronchodilator; pulmonary; genotype; pharmacogenomics; corticosteroid; allergy; immunology
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arg/Arg genotype on Advair (Fluticasone with Salmeterol) HFA (Active Comparator): Asthma patients with the Arg/Arg genotype who are randomized to continue the combination therapy of a specific long-acting beta 2 agonist (salmeterol) and inhaled corticosteroid (fluticasone) in the form of Advair HFA.
  Interventions: Drug: Fluticasone with salmeterol; Drug: Ipratropium HFA; Drug: Albuterol HFA
- Gly/Gly genotype on Advair (Fluticasone with Salmeterol) HFA (Active Comparator): Asthma patients with the Gly/Gly genotype who are randomized to continue the combination therapy of a specific long-acting beta 2 agonist (salmeterol) and inhaled corticosteroid (fluticasone) in the form of Advair HFA.
  Interventions: Drug: Fluticasone with salmeterol; Drug: Ipratropium HFA; Drug: Albuterol HFA
- Arg/Arg genotype on Fluticasone HFA (Experimental): Asthma patients with the Arg/Arg genotype who are randomized to fluticasone (Flovent HFA) alone.
  Interventions: Drug: Fluticasone HFA; Drug: Ipratropium HFA; Drug: Albuterol HFA
- Gly/Gly genotype on Fluticasone HFA (Experimental): Asthma patients with the Gly/Gly genotype who are randomized to fluticasone (Flovent HFA) alone.
  Interventions: Drug: Fluticasone HFA; Drug: Ipratropium HFA; Drug: Albuterol HFA

INTERVENTIONS:
Drug: Fluticasone with salmeterol — Fluticasone 45mcg, 115mcg, or 230mcg with salmeterol 21mcg, via HFA device, 2 puffs every 12 hrs, over 16 week study period.
  Other Names: Advair HFA
  Arms: Arg/Arg genotype on Advair (Fluticasone with Salmeterol) HFA; Gly/Gly genotype on Advair (Fluticasone with Salmeterol) HFA
Drug: Fluticasone HFA — Fluticasone HFA alone at 44mcg, 110mcg or 220 mcg 2 puffs every 12 hrs, over 16 week study period.
  Other Names: Flovent HFA
  Arms: Arg/Arg genotype on Fluticasone HFA; Gly/Gly genotype on Fluticasone HFA
Drug: Ipratropium HFA — Primary as-needed rescue medication in all treatment groups
  Other Names: Atrovent
Drug: Albuterol HFA — Secondary as-needed rescue medication in all treatment groups

SUMMARY:
The investigators are conducting a study of asthma patients who use fluticasone with salmeterol (Advair) or any other combination of an inhaled corticosteroid (ICS) and a long acting beta agonist (LABA) to manage their asthma symptoms.

Participants begin the study by continuing to use fluticasone with salmeterol or substituting fluticasone with salmeterol for their current ICS/LABA medication at their regular dose or the comparable dose(all study medications are provided) for a six-week period. Patients are then separated into 2 groups: one group is asked to use fluticasone (Flovent), the other to use fluticasone with salmeterol , twice daily over a 16-week period (patients will need to be seen monthly during this time). Neither study personnel nor patients will know which drug is being used.

Patients are also asked to use a peak flow meter and record their daily results on a form, along with the number of puffs they use of their rescue inhaler each day. They also record any changes in asthma medications and information on any asthma episodes.

The investigators hypothesize that there are certain patients with asthma who will do better when a long acting beta agonist is removed from their maintenance asthma medications.

DETAILED DESCRIPTION:
Beta 2 (b2) agonists are the most common type of bronchodilator used to treat asthma. Beta 2 (b2) agonists are agents that bind to b2 receptors and cause muscle relaxation of the airways. There are different variants of the gene (genotypes) that influence how b2 agonists perform among the population.

A recent study demonstrated that patients with mild asthma and the Arg/Arg variant at the 16th amino acid position have improved lung function and asthma control when albuterol (Proventil-HFA), a short acting b2 agonist, is replaced with a different class of bronchodilator. The investigators plan to study asthma patients with distinct genetic makeups of the b2 receptor; specifically Arg/Arg and Gly/Gly.

Throughout the treatment period, patients will be instructed to use ipratropium bromide (Atrovent-HFA), a bronchodilator which works through a different mechanism for rescue therapy; albuterol will be available for use if necessary.

The goal of this study is to determine if the withdrawal of a beta 2 agonist leads to improved asthma control in those asthmatic patients with the Arg/Arg genotype compared with those with the Gly/Gly genotype.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of moderate or severe and persistent asthma
* Currently being treated with a long acting beta agonist and inhaled corticosteroid
* Forced expiratory volume at one second (FEV1) > or = 70% at randomization visit (pulmonary function test result)
* Women of childbearing potential must be on an effective form of contraception
* Ability to read and understand English

Exclusion Criteria:

* Active smoking or greater than 10-pack-year history of smoking
* History of intubation for asthma within the past 10 years
* Patients who are pregnant, become pregnant during the study or are breast feeding
* Major comorbidity including: severe cardiac disease, uncontrolled hypertension, poorly controlled diabetes, malignancy within the past 5 years (except non-melanoma skin lesions), and pulmonary disease other than asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Slankard, M.D., Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center Eastside, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 90 participants enrolled (40 Arg/Arg Genotype and 50 Gly/Gly Genotype). Nine Arg/Arg participants and 14 Gly/Gly participants were not randomized due to dropout or ineligibility.
Period: Overall Study
Arm/Group | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA | Arg/Arg Genotype on Fluticasone HFA | Gly/Gly Genotype on Fluticasone HFA
Started | 15 | 18 | 16 | 18
Completed | 15 | 17 | 13 | 16
Not Completed | 0 | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA: Asthma patients with the Arg/Arg genotype who are randomized to continue the combination therapy of a specific long-acting beta 2 agonist (salmeterol) and inhaled corticosteroid (fluticasone) in the form of Advair HFA.
  Drug: Fluticasone with salmeterol Fluticasone 45mcg, 115mcg, or 230mcg with salmeterol 21mcg, via HFA device, 2 puffs every 12 hrs, over 16 week study period.
  Other Name: Advair HFA
  Drug: Ipratropium HFA Primary as-needed rescue medication in all treatment groups Other Name: Atrovent
  Drug: Albuterol HFA Secondary as-needed rescue medication in all treatment groups
- Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA: Asthma patients with the Gly/Gly genotype who are randomized to continue the combination therapy of a specific long-acting beta 2 agonist (salmeterol) and inhaled corticosteroid (fluticasone) in the form of Advair HFA.
  Drug: Fluticasone with salmeterol Fluticasone 45mcg, 115mcg, or 230mcg with salmeterol 21mcg, via HFA device, 2 puffs every 12 hrs, over 16 week study period.
  Other Name: Advair HFA
  Drug: Ipratropium HFA Primary as-needed rescue medication in all treatment groups Other Name: Atrovent
  Drug: Albuterol HFA Secondary as-needed rescue medication in all treatment groups
- Arg/Arg Genotype on Fluticasone HFA: Asthma patients with the Arg/Arg genotype who are randomized to fluticasone (Flovent HFA) alone.
  Drug: Fluticasone HFA Fluticasone HFA alone at 44mcg, 110mcg or 220 mcg 2 puffs every 12 hrs, over 16 week study period.
  Other Name: Flovent HFA
  Drug: Ipratropium HFA Primary as-needed rescue medication in all treatment groups Other Name: Atrovent
  Drug: Albuterol HFA Secondary as-needed rescue medication in all treatment groups
- Gly/Gly Genotype on Fluticasone HFA: Gly/Gly genotype on Fluticasone HFA
  Drug: Fluticasone HFA Fluticasone HFA alone at 44mcg, 110mcg or 220 mcg 2 puffs every 12 hrs, over 16 week study period.
  Other Name: Flovent HFA
  Drug: Ipratropium HFA Primary as-needed rescue medication in all treatment groups Other Name: Atrovent
  Drug: Albuterol HFA Secondary as-needed rescue medication in all treatment groups
- Total: Total of all reporting groups
Arm/Group | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA | Arg/Arg Genotype on Fluticasone HFA | Gly/Gly Genotype on Fluticasone HFA | Total
Number analyzed (Participants) | 15 | 17 | 13 | 16 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 13 | 16 | 61
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 12 | 12 | 47
  Male | 2 | 7 | 1 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 7 | 7 | 10 | 32
  African-American | 5 | 6 | 3 | 4 | 18
  Asian | 0 | 3 | 2 | 0 | 5
  Other | 2 | 1 | 1 | 2 | 6
  Hispanic | 1 | 3 | 3 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Morning Peak Flow
Description: Absolute change in morning peak flow at the end of the 16-week study period compared with baseline (last two weeks of run-in). Peak flow measurement is a test to measure air flowing out of the lung.
Time Frame: Up to 16 weeks from baseline
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA | Arg/Arg Genotype on Fluticasone HFA | Gly/Gly Genotype on Fluticasone HFA
Number analyzed (Participants) | 15 | 17 | 13 | 16
L/min | -15.7 (69.6) | 8.4 (29.7) | -5.6 (17.9) | -14.4 (36.2)

2. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) Pre-Bronchodilator
Description: Change in Forced Expiratory Volume in 1 Second (FEV1) Pre-Bronchodilator as measured by spirometry
Time Frame: Up to 16 weeks from baseline
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA | Arg/Arg Genotype on Fluticasone HFA | Gly/Gly Genotype on Fluticasone HFA
Number analyzed (Participants) | 15 | 17 | 13 | 16
Liter | -0.03 (0.20) | -0.08 (0.21) | -0.12 (0.16) | -0.11 (0.27)

3. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) Post-Bronchodilator
Description: Change in Forced Expiratory Volume in 1 Second (FEV1) Post-Bronchodilator as measured by spirometry
Time Frame: Up to 16 weeks from baseline
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA | Arg/Arg Genotype on Fluticasone HFA | Gly/Gly Genotype on Fluticasone HFA
Number analyzed (Participants) | 15 | 17 | 13 | 16
Liter | 0.02 (0.20) | -0.07 (0.19) | -0.11 (0.18) | -0.07 (0.17)

4. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) Percent Predicted Pre-Bronchodilator
Description: Change in Forced Expiratory Volume in 1 Second (FEV1) Percent Predicted Pre-Bronchodilator as measured by spirometry
Time Frame: Up to 16 weeks from baseline
Measure: Mean (Standard Deviation); unit: Percent Predicted
Arm/Group | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA | Arg/Arg Genotype on Fluticasone HFA | Gly/Gly Genotype on Fluticasone HFA
Number analyzed (Participants) | 15 | 17 | 13 | 16
Percent Predicted | -1.0 (7.6) | -2.5 (7.5) | -3.8 (5.5) | -3.3 (9.4)

5. Secondary Outcome: Change in Asthma Symptom Score
Description: Asthma symptom score measures asthma symptoms on a scale from 0 to 3. 0 = No asthma symptoms; 1 = 1-3 asthma episodes each lasting 2 hours or less, all mild; 2= 4 or more asthma episodes that interfered with activity, play, school, or sleep for less than 2 hours; 3= 1 or more asthma episodes lasting longer than 2 hours, or resulting in shortening normal activity, or seeing a doctor, or going to a hospital. A higher score indicates a worse outcome.
Time Frame: Up to 16 weeks from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA | Arg/Arg Genotype on Fluticasone HFA | Gly/Gly Genotype on Fluticasone HFA
Number analyzed (Participants) | 15 | 17 | 13 | 16
score on a scale | 0.3 (3.5) | -1.2 (3.2) | 0.4 (4.1) | 0.5 (1.2)

ADVERSE EVENTS:
Description: Adverse event data were collected and reported in the groups in which they were analyzed during the 16-week treatment period.
Arm/Group | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA | Arg/Arg Genotype on Fluticasone HFA | Gly/Gly Genotype on Fluticasone HFA
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 3/15 | 3/17 | 3/13 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arg/Arg Genotype on Advair (Fluticasone With Salmeterol) HFA (N=15) | Gly/Gly Genotype on Advair (Fluticasone With Salmeterol) HFA (N=17) | Arg/Arg Genotype on Fluticasone HFA (N=13) | Gly/Gly Genotype on Fluticasone HFA (N=16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Right Foot Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pharyngitis (General disorders) | 0 | 0 | 1 | 0
Gastric Reflux (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Wheeze (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Motor Vehicle Accident (General disorders) | 0 | 0 | 0 | 1
Compressed Cervical Nerve (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No